CLINICAL TRIAL: NCT02536846
Title: The Effects of Antipsychotic Drugs on Brain Metabolism in Healthy Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dost Ongur (Other)
Responsible Party: Sponsor-Investigator, Dost Ongur, Chief of Psychotic Disorders Division at McLean Hospital and Associate Professor in Psychiatry at Harvard Medical School, Mclean Hospital
Organization: Mclean Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015P001140; 041512 (Other Grant/Funding Number: McLean Hospital)
Record Dates: First submitted 2015-08-20; First posted 2015-09-01 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Healthy volunteers; antipsychotic drugs; brain metabolism
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Second Generation Antipsychotic Drug (Experimental): Olanzapine; a single 2.5 mg dose PO daily followed by 5 mg dose PO daily for 14 days
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — All subjects will take a single 2.5 mg dose of olanzapine (Zyprexa Zydis) followed by a 5 mg dose for 14 days. (2.5 mg/d for 1 day, 5 mg/d for 14 days).
  Other Names: Zyprexa Zydis 5 mg tb

SUMMARY:
The primary aim of this study is to investigate antipsychotic drug effects on healthy brain metabolism.

DETAILED DESCRIPTION:
Schizophrenia is a complex psychiatric disorder characterized by alterations in brain structure. It is not clear yet whether some of these alterations are primarily related to pathophysiology of illness per se or consequence of brain exposure to the effects of psychotropic drugs. In recent years accumulating evidence suggests that exposure to the effects of psychotropic drugs may contribute to the structural and other changes in brain. Therefore, use of antipsychotic medications as treatment for schizophrenia represents a potential confounding factor in many of the studies. Most neuroimaging studies of schizophrenia to date have not included the examination of non-medicated patients, making conclusions about medication effects on neuroimaging measures difficult. MRI studies of structural brain changes across time are limited by the fact that due to ethical reasons neither untreated subjects with schizophrenia nor control subjects exposed to antipsychotic medications can be used as comparison groups. There are some preclinical rat and primate models which revealed chronic antipsychotic-induced alterations in the brain. However few studies investigate the effects of chronic exposure to antipsychotic drugs on healthy human brain. Therefore in this study, investigators aimed to evaluate brain alterations induced by chronic drug exposure in healthy volunteers. To address this problem, we will conduct a single-site, single arm, open-label, interventional, multimodal neuroimaging study of healthy comparison subjects who are exposed to antipsychotic medication for 15 days. This study will include up to 40 healthy adult (21-50 years old) volunteers. Participants will be recruited via online advertisements and flyers as well as approaching healthy individuals who participated in previous studies. Investigators have three aims: 1. to study the levels of chemicals and kinetics of enzymes associated with cellular energy metabolism in brain before and after use of antipsychotic drug (using 1P MRS). 2. to collect data on the structure of the gray matter and white matter; resting state functional brain activity; levels of brain chemicals including glutamate and GABA; and white matter integrity before and after use of antipsychotic drug (using structural MRI, fMRI, dTI, 1H MRS). 3. to investigate side effects of antipsychotic drugs. It was planed to give healthy participants a single 2.5 mg dose of olanzapine followed by a 5 mg dose for 14 days. Olanzapine, a second generation antipsychotic agent, was selected to administer because this medication has strong effects on energy metabolism in general. The recommended daily dose range for olanzapine is indicated as 10-30 mg/d in the last "APA (American Psychiatric Association) Practice Guideline for the Treatment of Patients With Schizophrenia". A recent study suggests that minimum effective dose for olanzapine in schizophrenia is 7.5 mg/d (the upper range of 5 mg ± 2.5 mg/d) and higher olanzapine doses (10, 10 ± 2.5, 15, and 15 ± 2.5 mg/d) are more efficacious than placebo. Therefore it was determined to give healthy subjects only 5 mg/d olanzapine, the lower limit of the optimal dose range (5 mg ± 2.5 mg/d), to mimic the therapeutic effect but also protect the participants from adverse effects of treatment. As the goal is to examine the effects of chronic drug use, the duration of medication was determined to be 15 days, the longest but historically safe olanzapine usage period in healthy individuals up to now. There is no published literature on the effects of olanzapine on brain measures. Therefore, it is not possible to calculate a sample size that would detect a given between-group difference in this study. Investigators plan to recruit a sample that is large enough to establish the absence of a moderate or large effect. It was proposed that sample size of 30 subjects will be sufficient to detect a difference with effect sizes of 0.45 or greater as significant at the p<0.05 level with 80% power. Effect sizes of 0.5 are generally considered moderate and 0.8 considered large. Therefore, a not-statistically significant finding with this sample size will suggest that any effects of olanzapine on brain metabolism are small at most. Investigators will collect interview and neuroimaging data at baseline and after the medication period. Deviations induced by the study drug on healthy brain will be examined using paired t-tests for before and after measurements. Investigation of parameters before and after the use of antipsychotic drug in healthy people will give a chance to determine brain alterations related to drug itself, independent from the pathophysiology of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-50 years old
* Male or female
* Without psychiatric diagnosis according to a structured psychiatric interview (SCID)
* Without history of a psychotic disorder among parents, siblings, or children

Exclusion Criteria:

* Significant medical or neurological illness
* Diagnosis diabetes mellitus, uncontrolled hypertension, severe hypotension, coronary artery disease, metabolic syndrome, glaucoma, liver impairment, decreased renal function, respiratory disorders, peptic ulcer disease (absolute and relative contraindications to use of antipsychotic drugs)
* Body mass index (BMI) over 30
* Taking any other medications, including over the counter supplements with the exception of oral contraceptives for women
* Pregnancy. Females of child-bearing age must be using an effective contraceptive method
* History of smoking, substance abuse or dependence
* Contraindication to MR scan (claustrophobia, cardiac pacemakers, metal clips and stents on blood vessels, artificial heart valves, artificial arms, hands, legs, etc., brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings, other metallic surgical hardware in vital areas, certain tattoos with metallic ink, certain transdermal patches, metal-containing IUDs)
* Medical condition that would prevent blood draws

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Martinez ZA, Oostwegel J, Geyer MA, Ellison GD, Swerdlow NR. "Early" and "late" effects of sustained haloperidol on apomorphine- and phencyclidine-induced sensorimotor gating deficits. Neuropsychopharmacology. 2000 Nov;23(5):517-27. doi: 10.1016/S0893-133X(00)00147-0. PMID 11027917
- [Background] Agostinho FR, Reus GZ, Stringari RB, Ribeiro KF, Ferraro AK, Benedet J, Rochi N, Scaini G, Streck EL, Quevedo J. Treatment with olanzapine, fluoxetine and olanzapine/fluoxetine alters citrate synthase activity in rat brain. Neurosci Lett. 2011 Jan 10;487(3):278-81. doi: 10.1016/j.neulet.2010.10.037. Epub 2010 Oct 28. PMID 20971158
- [Background] Dorph-Petersen KA, Pierri JN, Perel JM, Sun Z, Sampson AR, Lewis DA. The influence of chronic exposure to antipsychotic medications on brain size before and after tissue fixation: a comparison of haloperidol and olanzapine in macaque monkeys. Neuropsychopharmacology. 2005 Sep;30(9):1649-61. doi: 10.1038/sj.npp.1300710. PMID 15756305
- [Background] Konopaske GT, Dorph-Petersen KA, Pierri JN, Wu Q, Sampson AR, Lewis DA. Effect of chronic exposure to antipsychotic medication on cell numbers in the parietal cortex of macaque monkeys. Neuropsychopharmacology. 2007 Jun;32(6):1216-23. doi: 10.1038/sj.npp.1301233. Epub 2006 Oct 25. PMID 17063154
- [Background] Konopaske GT, Dorph-Petersen KA, Sweet RA, Pierri JN, Zhang W, Sampson AR, Lewis DA. Effect of chronic antipsychotic exposure on astrocyte and oligodendrocyte numbers in macaque monkeys. Biol Psychiatry. 2008 Apr 15;63(8):759-65. doi: 10.1016/j.biopsych.2007.08.018. Epub 2007 Oct 22. PMID 17945195
- [Background] Vita A, De Peri L. The effects of antipsychotic treatment on cerebral structure and function in schizophrenia. Int Rev Psychiatry. 2007 Aug;19(4):429-36. doi: 10.1080/09540260701486332. PMID 17671875
- [Background] Smieskova R, Fusar-Poli P, Allen P, Bendfeldt K, Stieglitz RD, Drewe J, Radue EW, McGuire PK, Riecher-Rossler A, Borgwardt SJ. The effects of antipsychotics on the brain: what have we learnt from structural imaging of schizophrenia?--a systematic review. Curr Pharm Des. 2009;15(22):2535-49. doi: 10.2174/138161209788957456. PMID 19689326
- [Background] Leucht S, Samara M, Heres S, Patel MX, Woods SW, Davis JM. Dose equivalents for second-generation antipsychotics: the minimum effective dose method. Schizophr Bull. 2014 Mar;40(2):314-26. doi: 10.1093/schbul/sbu001. Epub 2014 Feb 3. PMID 24493852
- [Background] Vidarsdottir S, Roelfsema F, Frolich M, Pijl H. Olanzapine shifts the temporal relationship between the daily acrophase of serum prolactin and cortisol concentrations rhythm in healthy men. Psychoneuroendocrinology. 2009 Jun;34(5):705-12. doi: 10.1016/j.psyneuen.2008.11.008. Epub 2009 Jan 7. PMID 19131173
- [Background] Vidarsdottir S, de Leeuw van Weenen JE, Frolich M, Roelfsema F, Romijn JA, Pijl H. Effects of olanzapine and haloperidol on the metabolic status of healthy men. J Clin Endocrinol Metab. 2010 Jan;95(1):118-25. doi: 10.1210/jc.2008-1815. Epub 2009 Nov 11. PMID 19906788
- [Background] Sacher J, Mossaheb N, Spindelegger C, Klein N, Geiss-Granadia T, Sauermann R, Lackner E, Joukhadar C, Muller M, Kasper S. Effects of olanzapine and ziprasidone on glucose tolerance in healthy volunteers. Neuropsychopharmacology. 2008 Jun;33(7):1633-41. doi: 10.1038/sj.npp.1301541. Epub 2007 Aug 22. PMID 17712347
- [Background] Vidarsdottir S, Vlug P, Roelfsema F, Frolich M, Pijl H. Orally disintegrating and oral standard olanzapine tablets similarly elevate the homeostasis model assessment of insulin resistance index and plasma triglyceride levels in 12 healthy men: a randomized crossover study. J Clin Psychiatry. 2010 Sep;71(9):1205-11. doi: 10.4088/JCP.08m04654yel. Epub 2010 Apr 20. PMID 20441717
- [Background] Fountaine RJ, Taylor AE, Mancuso JP, Greenway FL, Byerley LO, Smith SR, Most MM, Fryburg DA. Increased food intake and energy expenditure following administration of olanzapine to healthy men. Obesity (Silver Spring). 2010 Aug;18(8):1646-51. doi: 10.1038/oby.2010.6. Epub 2010 Feb 4. PMID 20134408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals between 21-50 years old without a psychiatric or serious medical diagnosis or family history or first degree relative with a psychotic disorder.
Groups:
- Olanzapine: Participants will take olanzapine, Zyprexa Zydis, 5mg daily for 15 days.
Period: Overall Study
Arm/Group | Olanzapine
Started (35 participants were enrolled and 10 were allocated to receive olanzapine.) | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Individuals between 21-50 years old without a psychiatric or serious medical diagnosis or family history or first degree relative with a psychotic disorder.
Arm/Group | Second Generation Antipsychotic Drug
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.42 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Nicotinamide Adenine Dinucleotide Metabolites NAD+/NADH
Description: Change in brain nicotinamide adenine dinucleotide NAD+/NADH metabolite ratio as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Olanzapine
Number analyzed (Participants) | 7
ratio | -0.79 (2.37)

2. Primary Outcome: Change in Brain Phosphocreatine (PCr)
Description: Change in Phosphocreatine (PCr) metabolite concentration as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: Baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
ratio | 0.01 (0.11)

3. Primary Outcome: Change in Brain Creatine Kinase (CK) Forward Reaction Rate
Description: Change in forward reaction rate constant (kf) of the creatine kinase (CK) as measured by in vivo 31P magnetic resonance spectroscopy magnetization transfer
Time Frame: Baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: s-1
Arm/Group | Olanzapine
Number analyzed (Participants) | 4
s-1 | -0.04 (0.08)

4. Primary Outcome: Change in Brain Parenchymal pH
Description: Change in brain parenchymal pH as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
pH | 0.00 (0.01)

5. Secondary Outcome: Change in Volumes of the Frontal, Parietal and Temporal Lobe Regions
Description: Change in the gray matter volumes (cubic millimeters) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas. Data was acquired using structural magnetic resonance imaging (MRI) at 3T.
Time Frame: baseline and after 15 day medication period
Measure: Mean (Standard Deviation); unit: cubic mm
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
cubic mm
  Frontal Lobe | -2500.44 (4304.17)
  Parietal Lobe | -600 (1264.79)

6. Secondary Outcome: Change in Surface Area of the Frontal, Parietal and Temporal Regions
Description: Change in the cortical surface area (millimeters squared) of the frontal, parietal and temporal lobes as defined by Freesurfer's Desikan-Killiany Brain Atlas. Data was acquired using structural magnetic resonance imaging (MRI) at 3T.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
mm^2
  Frontal lobe | -801.19 (1563.02)
  Parietal lobe | -581.56 (1272.93)

7. Secondary Outcome: Change in fMRI Resting State Functional Connectivity
Description: Change in resting state functional connectivity to the medial prefrontal cortex and superior parietal lobules following olanzapine administration period. Whole-brain, seed-to-voxel analyses were conducted utilizing anatomically-defined seed regions and age-corrected within-subjects f-tests were run to determine the presence and size (in voxels) of clusters where connectivity changed significantly following olanzapine administration. Results are reported in units of voxels for each cluster meeting a threshold of voxel-level uncorrected p<.001 and cluster-level p-FDR<.05. A result of zero indicates that no clusters were identified within subjects as changed in connectivity relative to the seed regions.
Time Frame: baseline and after 15 days medication period
Population: Number of voxels that showed significant change in connectivity following administration of olanzapine.
Measure: Number; unit: Voxels
Arm/Group | Olanzapine
Number analyzed (Participants) | 7
Voxels
  medial prefrontal cortex | 0
  superior parietal lobule | 0

8. Secondary Outcome: Change in GABA Concentration
Description: Change in GABA concentration measured by proton magnetic resonance spectroscopy.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
mmol | 0.11 (0.20)

9. Secondary Outcome: Change in Fractional Anisotropy (FA) Measured by Diffusion Tensor Imaging (DTI)
Description: Change in fractional anisotropy (FA), a scalar measure of diffusivity, of water in the brain assessed by DTI at 3T. FA values range from 0 (isotropic, meaning diffusion is equally restricted in 3D space) to 1 (anisotrophic, meaning that diffusion is completely restricted to a single direction).
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
Units on a scale
  Core FA | 0.0007 (0.01)
  Genu of corpus callosum | -0.003 (0.013)
  Cingulum | -0.008 (0.027)
  Inferior fronto-occipital fasciculus | -0.002 (0.012)
  Anterior thalamic radiation | 0.002 (0.015)

10. Secondary Outcome: Change in Glutamate Metabolite Concentration
Description: Change in glutamate metabolite concentration measured by proton magnetic resonance spectroscopy.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: millimoles
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
millimoles | 0.13 (0.66)

11. Secondary Outcome: Change in MATRICS Cognitive Consensus Battery (MCCB) Total Composite Score
Description: Change in the MATRICS Cognitive Consensus Battery (MCCB), that includes 10 tasks that measure processing speed (Brief Assessment of Cognition in Schizophrenia - Symbol Coding, Animal Fluency, Trails A), attention (Continuous Performance Test), working memory (WMS-III Spatial Span, Letter-Number Span), verbal learning (Hopkins Verbal Learning Test - Revised), visual learning (Brief Visuospatial Memory Test - Revised), problem solving (Neuropsychological Assessment Battery Mazes) and social cognition (Mayer-Salovey-Caruso Emotional Intelligence Test). Scores from each subtest are normed and their T-scores are summed to yield a MCCB composite score, then the total composite T-score is standardized to normative data among a healthy population. The composite T-score has a mean of 50 and a standard deviation of 10. Higher total composite scores indicate better cognitive outcomes.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
Score on a scale | 3.63 (4.72)

12. Other Pre Specified Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: Change in Montgomery-Asberg Depression Rating Scale (MADRS) score, a 0-60 point scale rating depressive symptoms. Higher scores indicate more severe clinical symptoms.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.88 (3.00)

13. Other Pre Specified Outcome: Change in Beck Depression Inventory (BDI) Score
Description: Change in Beck Depression Inventory (BDI) score, a self-report questionnaire measuring depressive symptoms on a scale of 0-63. Scores ranging 0-9 generally indicate minimal depressive symptoms, while scores 10-18 indicate mild, 19-29 indicates moderate, and 30-63 indicates severe depressive symptoms, respectively.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.63 (1.30)

14. Other Pre Specified Outcome: Change in Young Mania Rating Scale (YMRS) Score
Description: Change in Young Mania Rating Scale (YMRS) score, an interview-based, 11-item scale that measures the severity of core features of clinical mania. 7 items are scored on a 0-4 point scale, while the remaining 4 are scored on a 0-8 point scale, for a total possible range of 0-64. Higher scores indicate more severe manic symptoms.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.875 (1.126)

15. Other Pre Specified Outcome: Change in Beck Anxiety Inventory (BAI) Score
Description: Change in Beck Anxiety Inventory (BAI) score, a self-report measure of anxiety symptoms. Scores range from 0-63, with higher scores indicating more severe anxiety.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.63 (1.41)

16. Other Pre Specified Outcome: Change in The Columbia Suicide Severity Rating Scale Score
Description: Change in The Columbia Suicide Severity Rating Scale score, a self-report scale measuring suicidality. Only the total score, not subscale of suicidal ideation intensity, will be measured. Total scores can range from 0-10, with higher scores indicating increased suicidality.
Time Frame: baseline and 2, 5, 10, 15 days during medication period
Population: Data for this measure was collected for 10 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Generation Antipsychotic Drug
Number analyzed (Participants) | 10
score on a scale
  Baseline | 0 (0)
  After 2 days medication | 0 (0)
  After 5 days medication: number analyzed (Participants) | 9
  After 5 days medication | 0 (0)
  After 10 days medication: number analyzed (Participants) | 9
  After 10 days medication | 0 (0)
  After 15 days medication: number analyzed (Participants) | 9
  After 15 days medication | 0 (0)

17. Other Pre Specified Outcome: Change in Pittsburgh Sleep Quality Index Score
Description: Change in Pittsburgh Sleep Quality Index score, a measurement of sleep quality. The index measures 7 sleep components on a 0-3 scale; each of the 7 raw scores is summed to get a global score. The global score ranges from 0-21, with higher scores indicating poor sleep quality. Scores >5 are typically considered poor sleep quality.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.63 (1.92)

18. Other Pre Specified Outcome: Change in LUNSERS (Liverpool University Neuroleptic Side Effect Rating Scale) Score
Description: Change in LUNSERS (Liverpool University Neuroleptic Side Effect Rating Scale) score, a self-report measure of antipsychotic side effects. The scale has 51 questions, 41 of which are about side-effects and 10 "red herrings" for validation purposes. The total neuroleptic side effect score is derived from the sum of the 41 side-effect questions, with a potential range of 0-164. Higher scores indicate more severe neuroleptic side effects.
Time Frame: baseline and 2, 5, 10 and 15 days (or final assessment) during medication period
Population: Data for this measure was collected for 10 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 10
score on a scale
  Baseline | 0.20 (0.63)
  2 days | 4.50 (4.99)
  5 days: number analyzed (Participants) | 9
  5 days | 2.11 (3.02)
  10 days: number analyzed (Participants) | 9
  10 days | 2.22 (3.19)
  Endpoint: number analyzed (Participants) | 8
  Endpoint | 3.90 (4.98)

19. Other Pre Specified Outcome: Change in Body Weight
Description: Change in participant body weight in kg, as measured using a standing scale.
Time Frame: baseline and 2, 5, 10 and 15 days (or final assessment) during medication period
Population: Data for this measure was collected for 10 participants
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Olanzapine
Number analyzed (Participants) | 10
kg
  Baseline | 0 (0)
  2 days | -0.29 (1.13)
  5 days: number analyzed (Participants) | 9
  5 days | 0.12 (1.41)
  10 days: number analyzed (Participants) | 9
  10 days | 0.21 (0.88)
  Endpoint | 0.73 (1.34)

20. Other Pre Specified Outcome: Change in Hip Circumference
Description: Change in the hip circumference measurement, taken as an average of 3 measures by tape measure
Time Frame: baseline and 2, 5, 10 and 15 days (or final assessment) during medication period
Population: Data for this measure was collected for 10 participants.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Olanzapine
Number analyzed (Participants) | 10
cm
  Baseline | 0 (0)
  2 days: number analyzed (Participants) | 9
  2 days | -0.43 (3.10)
  5 days: number analyzed (Participants) | 7
  5 days | -1.10 (4.27)
  10 days: number analyzed (Participants) | 9
  10 days | -1.62 (4.89)
  Endpoint | -1.24 (3.54)

21. Other Pre Specified Outcome: Change in Waist Circumference
Description: Change in waist circumference measurements, taken as an average of 3 measures by tape measure.
Time Frame: baseline and 2, 5, 10 and 15 days (or final assessment) during medication period
Population: Data was collected for 10 participants
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Olanzapine
Number analyzed (Participants) | 10
cm
  Baseline | 0 (0)
  After 2 days medication: number analyzed (Participants) | 9
  After 2 days medication | -0.47 (3.21)
  After 5 days medication: number analyzed (Participants) | 7
  After 5 days medication | 0.22 (1.36)
  After 10 days medication: number analyzed (Participants) | 9
  After 10 days medication | -0.23 (3.30)
  Endpoint | -0.15 (3.06)

22. Other Pre Specified Outcome: Change in Blood Glucose Levels
Description: Change in fasting serum glucose levels.
Time Frame: baseline and after 15 days during medication period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
mg/dL | 0.75 (6.18)

23. Other Pre Specified Outcome: Change in Fasting Total Cholesterol Level
Description: Change in fasting total cholesterol level
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
mg/dL | -1.75 (28.23)

24. Other Pre Specified Outcome: Change in Hemoglobin A1c Level
Description: Change in fasting, Hemoglobin A1c level
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
mmol/mol | -0.01 (0.11)

25. Other Pre Specified Outcome: Change in Serum Insulin Levels
Description: Change in insulin fasting serum levels
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
uIU/mL | -0.94 (1.73)

26. Other Pre Specified Outcome: Change in Prolactin Levels
Description: Change prolactin serum levels
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
ng/mL | 11.77 (20.69)

27. Other Pre Specified Outcome: Change in Total Caloric Intake
Description: Change in total caloric intake as assessed by the ASA24 Dietary Recall and Food Frequency Questionnaire - Revised. The ASA24 is a self-administered 24-hour dietary recall assessment.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Olanzapine
Number analyzed (Participants) | 7
kcal | 151.94 (1180.23)

28. Other Pre Specified Outcome: Change in The Wisconsin Schizotypy Scales - Short Form Scores
Description: Change in Wisconsin Schizotypy Scales (WSS) Short Form score, a self-report questionnaire assessing schizotypy in clinical and non-clinical samples. The measure has four scales, each with 15 True/False questions. There are 13 red-herring questions, that, if answered "True" invalidate the test. Each "false" response is scored 0, and each "true" response is scored 1. Scores for each scale range from 0 - 15, with higher scores indicating greater schizotypy. The WSS positive schizotypy score consists of the summed score of the perceptual aberration and magical ideation scales and scores range from 0-30, with higher scores indicating greater positive schizotypy. The WSS negative schizotypy score sums scores from the physical anhedonia and social anhedonia scales and ranges from 0-30, with higher scores indicating greater negative schizotypy.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale
  Change in positive schizotypy subscales | 0.06 (0.12)
  Change in negative schizotypy subscales | 0.09 (0.42)

29. Other Pre Specified Outcome: Change in the Early Psychosis Social Scale Survey Score
Description: Change in the Early Psychosis Social Scale score item of missed absences from school or work. Scores range from 1-5, with higher scores indicating more absences from school or work.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale | -0.13 (0.35)

30. Other Pre Specified Outcome: Change in the Prodromal Questionnaire, Brief Version Total Score
Description: Change in the Prodromal Questionnaire, Brief Version score, a 21 item self-report questionnaire designed to help identify those at ultra-high risk for developing psychotic symptoms. The total score is derived as the sum of all 21 items, with a possible range of 0-21. Higher scores indicate greater psychopathology.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 7
score on a scale | 0 (0)

31. Other Pre Specified Outcome: Change in the Symptoms Checklist - 90 - Revised Global Severity Score
Description: Changes in the Symptoms Checklist - 90 - Revised scale, which measures 9 domains of psychological dysfunction, summing to create an overall psychological distress (Global Severity Score). The scores of each of the 9 domains - somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism - combine for a total of 90 items, each measured on a 5-point scale. The sums of all 90 item scores, ranging 0-360, creates the Global Severity score. Higher scores indicate greater psychopathology.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 9
score on a scale | -2.33 (5.66)

32. Other Pre Specified Outcome: Change in the State-Trait Anxiety Inventory for Adults Scores
Description: Change in the State-Trait Anxiety Inventory for Adults, which measures both state and trait anxiety using 2 subscales for a total of 40 items. Each subscale has a range of 20-80, with higher scores indicating greater state or trait anxiety, respectively.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale
  Change in State-anxiety scale | -0.25 (2.38)
  Change in Trait-anxiety scale | -0.75 (2.38)

33. Other Pre Specified Outcome: Change in the World Health Organization Quality of Life Questionnaire Score
Description: Change in the World Health Organization Quality of Life questionnaire score, a 26-item assessment of overall quality of life. The questionnaire encompasses 4 domains: physical health, psychological health, social relationships, and environment. There are two additional questions, which assess the participant's perceptions of their own quality of life and physical health. Higher scores indicate better quality of life. Scores are summed within each domain. Total score is obtained by transforming for a total range of 0-100 within each domain.
Time Frame: baseline and after 15 days medication period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 8
score on a scale
  Change in physical health score | 2.25 (7.61)
  Change in psychological health score | -4.38 (7.25)
  Change in social relationships score | 0.75 (3.85)
  Change in environment score | -7.875 (12.15)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at all scheduled visits throughout the 15 day medication period at days 1, 2, 5, 10, and 15.
Arm/Group | Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=10)
Drowsiness (Nervous system disorders) | 10 (10)
Difficulty staying awake (Nervous system disorders) | 5 (5)
Sleeping too much (Nervous system disorders) | 4 (4)
Increased lipids (Metabolism and nutrition disorders) | 3 (3)
Increased food cravings (Metabolism and nutrition disorders) | 3 (3)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Vivid dreaming (Psychiatric disorders) | 2 (2)
Elevated LFTs (Hepatobiliary disorders) | 2 (2)
Difficulty getting to sleep (Psychiatric disorders) | 2 (2)
Shakiness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Increased thirst (General disorders) | 2 (2)
Elevated prolactin (Endocrine disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Slowing of movements (General disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT02536846/Prot_SAP_000.pdf